CLINICAL TRIAL: NCT06707324
Title: Analgesic Efficacy of Transversus Abdominis Plane Block Versus External Oblique Block in Patients Undergoing Elective Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2024-201012
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Transversus Abdominis Plane Block; External Oblique Block; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAB group (Active Comparator): 20 ml of 0.25% bupivacaine + 8 mg dexamethasone between the rectus abdominis muscle and the transversus abdominis muscle on both sides
  Interventions: Procedure: drug injected between the rectus abdominis muscle and the transversus abdominis muscle
- EOB group (Active Comparator): 20 ml of 0.25% bupivacaine+ 8 mg dexamethasone into the external oblique intercostal plane on both sides
  Interventions: Procedure: drug injected in the external oblique intercostal plane on both sides

INTERVENTIONS:
Procedure: drug injected between the rectus abdominis muscle and the transversus abdominis muscle — 20 ml of 0.25% bupivacaine + 8 mg dexamethasone between the rectus abdominis muscle and the transversus abdominis muscle on both sides
  Arms: TAB group
Procedure: drug injected in the external oblique intercostal plane on both sides — 20 ml of 0.25% bupivacaine+ 8 mg dexamethasone into the external oblique intercostal plane on both sides
  Arms: EOB group

SUMMARY:
Postoperative pain management is a critical aspect of recovery following laparoscopic cholecystectomy, a commonly performed procedure for symptomatic gallbladder disease. Effective analgesia not only enhances patient comfort but also facilitates early mobilization, reduces the incidence of complications, and improves overall outcomes.

Oblique subcostal transversus abdominis plane block (OSTAP), one of the regional anesthesia techniques, is used in middle and upper abdominal surgeries OSTAP blocks the T6-9 intercostal nerves between the rectus abdominis and transversus abdominis muscle. Many studies have shown that OSTAP block reduces the postoperative analgesic and opioid requirement and improves the quality of postoperative pain control.

DETAILED DESCRIPTION:
the potential mechanism of the external oblique intercostal fascial plane block (EOIB) in a cadaver study in which both lateral and anterior branches of the intercostal nerves T7-T10 were stained. Patients to whom this block was applied exhibited consistent dermatomal sensory blockade between T6-T10 in the anterior axillary line and T6-T9 in the midline. It has been shown that this block can be used in the clinical setting for upper abdominal wall analgesia.

Various adjuvants have been used to improve the quality and increase the duration of the local anesthetic action in different peripheral nerves and regional block techniques. dexamethasone microspheres have increased the block duration in both human and animal studies. Furthermore, dexamethasone has been shown to possess antiinflamatory action.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-60 years.
2. Gender: Both males and females.
3. BMI less than 35 kg/m2
4. Scheduled for laparoscopic cholecystectomy surgery
5. American Society of Anesthesiologists - ASA - I & II

Exclusion Criteria:

1-ASA physical status more than II. 2-History of allergic response to local anaesthetics or any of the medications used in the study

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
the first analgesic request depending on Numeric Rating Scale | 24hours
  the first analgesic request depending on Numeric Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut University, Assiut, Egypt,, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Result] Wang W, Wang L, Gao Y. A Meta-Analysis of Randomized Controlled Trials Concerning the Efficacy of Transversus Abdominis Plane Block for Pain Control After Laparoscopic Cholecystectomy. Front Surg. 2021 Aug 4;8:700318. doi: 10.3389/fsurg.2021.700318. eCollection 2021. PMID 34422893